CLINICAL TRIAL: NCT03108768
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2016_37
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2016_37
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Hearing Loss, Bilateral Sensorineural, Progressive
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Phonak Virto V and the successor of Phonak Virto V will be fitted to the participants individual hearing loss.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successor of Phonak Virto V (Experimental): The successor of Phonak's Virto V will be fitted to the participants individual hearing loss.
  Interventions: Device: Hearing Aid (Successor of Phonak Virto V)
- Phonak Virto V (Active Comparator): Phonak Virto V will be fitted to the participants individual hearing loss.
  Interventions: Device: Hearing Aid (Phonak Virto V)

INTERVENTIONS:
Device: Hearing Aid (Successor of Phonak Virto V) — The successor of Phonak's In-The-Ear (ITE) hearing aid Virto V will be fitted to the participants individual hearing loss.
  Arms: Successor of Phonak Virto V
Device: Hearing Aid (Phonak Virto V) — Phonak's In-The-Ear (ITE) hearing aid Virto V will be fitted to the participants individual hearing loss.
  Arms: Phonak Virto V

SUMMARY:
A methodical evaluation of new CE-labelled Phonak Hearing Systems is intended to be conducted on hard of participants with a hearing loss to grant quality control prior to product launch. The aim of the investigation series is to ensure zero-defect overall performance of the new hearing systems as well as maximum benefit for the participant with the devices in comparison to previously outstanding Phonak Hearing Systems.

DETAILED DESCRIPTION:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials in the way as planned for this study ("phase of final inspection"). This will be a controlled, single blinded and randomised active comparator clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years) with and without (experience with) hearing aids
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility in noise as signal to noise ratio in dB (dB SNR) | Three weeks
  The data, serving as primary outcomes are collected in a series of lab appointments. The speech intelligibility in noise will be assessed with the aid of the german Oldenburg sentence test. The result is the signal to noise ratio in dB (dB SNR). Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.

SECONDARY OUTCOMES:
Speech intelligibility in percent in a quiet listening situation | One week
  The data, serving as secondary outcomes are collected in a series of lab appointments. The speech intelligibility in quiet will be assessed with the aid of the german rhyme test "Einsilber-Reimtest nach von Wallenberg und Kollmeier" (WaKo). The result is the speech intelligibility in percent. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Zero-defect performance in daily life | Three weeks
  The data, serving as secondary outcomes are collected in a series of home trials taking place between the lab trial appointments. The zero-defect performance in daily life (that means: no interruptions, distortions, artefacts, feedback, system noise or other malfunctions) will be assessed with the aid of quantitative questionnaires. The results are "Yes/No" replies and open-ended.

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No